CLINICAL TRIAL: NCT00006319
Title: Molecular and Clinical Studies of Primary Immunodeficiency Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000209; 00-HG-0209
Record Dates: First submitted 2000-09-30; First posted 2000-10-02 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2023-10-13

CONDITIONS: Wiskott- Aldrich Syndrome; ADA Deficient SCID
Keywords: X-Linked Agammagloblinemia; Wiskott-Aldrich Syndrome; Jak-3 SCID; X-Linked SCID; X-Linked Hyper-IgM Syndrome; Natural History
MeSH Terms: conditions — Wiskott-Aldrich Syndrome; X-Linked Combined Immunodeficiency Diseases; Hyper-IgM Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADA deficient SCID: Patients with ADA deficient SCID
- Wiskott-Aldrich syndrome: Male patients with Wiskott-Aldrich syndrome

SUMMARY:
This study will try to identify mutations in the genes responsible for primary immunodeficiency disorders (inherited diseases of the immune system) and evaluate the course of these diseases in patients over time to learn more about the medical problems they cause. The immune system is composed of various cells (e.g., T and B cells and phagocytes) and other substances (complement system) that protect the body from infections and cancer. Abnormalities in the gene(s) responsible for the function of these components can lead to serious infections and other immune problems.

Patients with Wiskott-Aldrich syndrome, adenosine deaminase (ADA) deficiency. Participants will undergo a medical and family history, physical examination, and additional procedures and tests that may include the following:

1. Blood tests for: routine laboratory studies (i.e. cell counts, enzyme levels, electrolytes, etc.); HIV testing; immune response to various substances; genetic testing; and establishment of cell lines to maintain a supply of cells for continued study
2. Urine and saliva tests for biochemical studies
3. Skin tests to assess response to antigens such as the viruses and bacteria responsible for tetanus, candida, tuberculosis, diphtheria, chicken pox, and other diseases.
4. Skin and lymph node biopsies for tissue and DNA studies
5. Chest X-ray, CT scans, or both to look for cancer or various infections.
6. Pulmonary function test to assess lung capacity and a breath test to test for H. pylori infection.
7. Dental, skin and eye examinations.
8. Treatment with intravenous immunoglobulins or antibodies to prevent infections.
9. Apheresis for collecting white blood cells to study cell function. In this procedure, whole blood is collected through a needle placed in an arm vein. The blood circulates through a machine that separates it into its components. The white cells are then removed, and the red cells, platelets and plasma are returned to the body, either through the same needle or through a second needle placed in the other arm.
10. Bone marrow sampling to study the disease. A small amount of marrow from the hipbone is drawn (aspirated) through a needle. The procedure can be done under local anesthesia or light sedation.
11. Placental and umbilical cord blood studies, if cord blood is available, to study stem cells (cells that form blood cells).

Information gained from this study may provide a better understanding of primary immunodeficiencies, leading to better diagnosis and treatment. In addition, study participants may receive medical and genetic counseling and may be found eligible for other NIH studies on these diseases.

DETAILED DESCRIPTION:
The purpose of this protocol is to study patients with primary immunodeficiency disorders with the goal of contributing to both the clinical and molecular understanding of this heterogeneous group of inherited diseases. Clinical issues to be addressed will include disease manifestations and evolution, as well prevention and management of medical problems. Patients with diseases of known molecular basis (including Wiskott-Aldrich syndrome, ADA deficiency, JAK3 deficiency and other syndromes) will be genotyped in order to investigate phenotype-genotype correlation. Patients with disease of unknown or incomplete genetic characterization will be studied with hopes of contributing to the identification of specific genes responsible for disease. Studies of fresh cells, cell lines and tissue samples will be performed to help characterize the patient s syndrome as well as to test the efficacy of genetic correction when available.

The outcome we seek is to improve our knowledge of the molecular basis, clinical presentation and evolution of primary immunodeficiency diseases and to collaborate to maintain or improve the health status of our patients. No investigational clinical interventions are planned under this protocol. It is anticipated that additional protocols will be generated from preliminary data gathered in this umbrella study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with a clinical history or signs and symptoms suggestive of a primary immune deficiency syndrome and their family members are eligible for inclusion in this study and they may be referred by their physician or self-referred. If possible, a local physician/clinical immunologist will be identified for self-referred patients to serve as primary reference. If screening of the patients, either by phone interview or review of their medical records indicates that the patient may have a primary immunodeficiency syndrome and is HIV-negative, the patient will be invited to come to the NIH and sign an informed consent. If family history is positive for immunodeficiency, the patients or family members may be asked to invite other relatives to contact the PI to participate in the study.

Patients who were enrolled under such inclusion criteria may continue to be seen under the protocol under the medical advisory supervision of Dr. Harry Malech. New enrollments will be limited to children with established and verified diagnosis of ADA-SCID cared for by our collaborators at UCLA and from whom we will only

receive blood samples.

EXCLUSION CRITERIA:

Inability of the subject or the subject s parent/guardian to provide informed consent.

Patients infected with the Human Immunodeficiency Virus before enrollment.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male patients with Wiskott-Aldrich syndrome and patients with ADA deficient SCID@@@
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2000-10-25 (Actual)

PRIMARY OUTCOMES:
To broaden our current knowledge of the molecular basis, clinical presentation, evolution and outcome of primary immunodeficiencydiseases. | Ongoing
  to broaden our current knowledge of the molecular basis, clinical presentation, evolution and outcome of primary immunodeficiencydiseases.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth K Garabedian, R.N., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Sokolic R, Maric I, Kesserwan C, Garabedian E, Hanson IC, Dodds M, Buckley R, Issekutz AC, Kamani N, Shaw K, Tan B, Bali P, Hershfield MS, Kohn DB, Wayne AS, Candotti F. Myeloid dysplasia and bone marrow hypocellularity in adenosine deaminase-deficient severe combined immune deficiency. Blood. 2011 Sep 8;118(10):2688-94. doi: 10.1182/blood-2011-01-329359. Epub 2011 Jul 1. PMID 21725047
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2000-HG-0209.html